CLINICAL TRIAL: NCT06737523
Title: A Multicenter, Prospective, Single-arm Clinical Study of Chiglitazar Sodium Combined With Venetoclax and Azacitidine (CVA) for the Treatment of Refractory/Relapsed Acute Myeloid Leukemia (R/R AML)
Brief Title: Chiglitazar Sodium Combined With Venetoclax and Azacitidine (CVA) for the Treatment of R/R AML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Bing, Xu, Principal Investigator, The First Affiliated Hospital of Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMDYYYXYK-15
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Acute Myeloid Leukemia; Relapse; Refractory AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CVA (Experimental): Chiglitazar Sodium in combination with Venetoclax and Azacitidine
  Interventions: Drug: CVA

INTERVENTIONS:
Drug: CVA — Chiglitazar Sodium in combination with Venetoclax and Azacitidine

SUMMARY:
To investigate the safety and efficacy of the CVA regimen, composed of Chiglitazar Sodium in combination with Venetoclax and Azacitidine, in the treatment of patients with refractory/relapsed acute myeloid leukemia (R/R AML).

DETAILED DESCRIPTION:
1. Sogletanib 48mg per dose, once daily; Venetoclax 400mg per dose, once daily for 4 weeks; Azacitidine 100mg, once daily, days 1-7. 28 days/cycle, at least 2 cycles.
2. The drug concentration of Venetoclax will be tested one week after oral administration, and the dose will be adjusted according to the concentration.
3. After 2 treatment courses, patients with stable disease (SD) or progressive disease (PD) may receive up to 1-2 additional courses. If the disease still shows no improvement, they will be withdrawn from the clinical study and other treatment options will be considered, including allogeneic hematopoietic stem cell transplantation.

Note: In special circumstances based on the patient's condition, laboratory test indicators, and adverse reactions, etc.; for Venetoclax dosage, if the white blood cell count is >25×10^9/L before administration, hydroxyurea may be given first to reduce the count to less than 25×10^9/L before adding Venetoclax, and then the concentration of Venetoclax will be tested and the dose adjusted according to the concentration.

ELIGIBILITY:
Inclusion Criteria:

1. Acute myeloid leukemia (AML) confirmed by histology. Relapsed or refractory AML, including: a) Refractory disease is defined as no remission after at least one prior treatment. b) Disease relapse is defined as 5% or more blasts in the bone marrow after remission. c) Patients with AML arising from myelodysplastic syndromes (including CMML) or myeloproliferative neoplasms (secondary AML, t-AML) are also eligible;
2. Age ≥18 years, male or female, with an expected survival of more than 3 months;
3. Estimated creatinine clearance ≥ 50 mL/min;
4. AST and ALT ≤ 3.0 x ULN (unless considered due to leukemia organ involvement), bilirubin ≤ 3.0 x ULN (unless considered due to leukemia organ involvement);
5. ECOG ≤ 2;
6. Subjects are non-pregnant or using contraceptive measures during treatment;
7. Capable of understanding and voluntarily providing informed consent.

Exclusion Criteria:

1. Acute promyelocytic leukemia (APL);
2. Active central nervous system leukemia;
3. Patients with clinically significant QTc interval prolongation (males > 450 ms; females > 470 ms), ventricular tachycardia and atrial fibrillation, second-degree heart block, history of myocardial infarction and congestive heart failure within the year prior to enrollment, and patients with clinically symptomatic coronary heart disease requiring medication;
4. Active, uncontrolled severe infection;
5. Other non-myeloid malignancies within the past 2 years;
6. Mental disorders that would impede study participation;
7. Previous solid organ transplantation (pre-treatment with SCT is allowed, but not allowed if the patient has GVHD or is still receiving immunosuppressive/GVHD treatment);
8. Any other conditions that, in the opinion of the investigator, make the patient unsuitable to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate (CR) | Up to 36 months
  The absolute neutrophil count is ≥1.0 × 10^3/μL, the platelet count is ≥1.0 × 10^5/μL, independent of red blood cell transfusions, and the percentage of bone marrow blasts is <5%. There are no circulating bone marrow blasts and blasts with Auer rods in the peripheral blood; no extramedullary disease is present.
Complete Remission with Incomplete Count Recovery (CRi) | Up to 36 months
  Meeting all CR criteria except for residual neutropenia <1.0 × 10^3/μL (1000/μL) or thrombocytopenia <1.0 × 10^5/μL (100,000/μL). Dependence on red blood cell (RBC) transfusions is also defined as CRi.
Partial remission rate (PR) | Up to 36 months
  Meets all hematological criteria for CR, but the percentage of blasts in the bone marrow aspirate sample has decreased by at least 50%, reaching between 5% and 25%.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Xu, Principal Investigator — The First Aiffiliated hosptical of xiamen University
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No